CLINICAL TRIAL: NCT06155903
Title: Peripheral Nerve Blocks vs Selective Spinal Anesthesia in Patients With Femur Fracture: A Prospective Randomized Controlled Study
Brief Title: Peripheral Nerve Blocks vs Selective Spinal Anesthesia in Patients With Femur Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Coviello, Researcher, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2-2023-533
Record Dates: First submitted 2023-07-02; First posted 2023-12-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Femur Fracture; Peripheral Nerve Block; Spinal Anesthesia
Keywords: SPINAL ANESTHESIA; FEMUR FRACTURE; NERVE BLOCK; LOCOREGIONAL ANESTHESIA
MeSH Terms: conditions — Femoral Fractures | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The triple-blind approach (operating room anesthetist, surgeon, and patient) will be implemented as follows: a team will prepare the anesthetic mixtures in a dedicated room, isolated from the operating room and the Post-Anesthesia Care Unit (PACU) where a different team will be then responsible for the intra and postoperative management. The surgery will be conducted by the surgeon and the surgical team without knowledge of the anesthesiology procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Spinal Anesthesia (Active Comparator): The participant will receive selective spinal anesthesia.
  Interventions: Procedure: Selective Spinal Anesthesia; Drug: Anesthesiological mixtures (Spinal anesthesia)
- Peripheral nerve blocks (Active Comparator): The participant will receive a combination of femoral nerve block, sciatic nerve block with parasacral approach, lateral femoral cutaneous nerve block and obturator nerve block.
  Interventions: Procedure: Peripheral nerve blocks; Drug: Anesthesiological mixtures (Peripheral nerve block)

INTERVENTIONS:
Procedure: Selective Spinal Anesthesia — Selective Spinal Anesthesia will be performed at the L2-L3 or L3-L4 interspace with the patients lying in the lateral position (fractured side up). Anesthesiologists will determine the needling point for spinal anesthesia with reference to Tuffier's line, a virtual line connecting the tops of the iliac crests of a patient. A small dose of LA (4 ml of 1% lidocaine) will be injected into the skin and soft tissues at the planned site of spinal needle insertion. The correct path for spinal needle placement will be identified with the needle infiltration. The technique will be performed aseptically in the subarachnoid space after observing clear Cephalo-Spinal Fluid (CSF) in the spinal needle 25 Gauge, and without releasing the CSF. Selected patients will receive Hypobaric Bupivacaine 0.5% 7.5 mg and Sufentanil 5 µg and will maintain the lateral position for 15 min. At the end of these they will be gently placed in supine position.
  Arms: Selective Spinal Anesthesia
Procedure: Peripheral nerve blocks — In this group, four nerve blocks will be associated to ensure adequate anesthesia and analgesia during surgery.
  Sciatic nerve blocks with para sacral approach will be performed with a needle connected to an electrical nerve stimulation. The needle will be advanced until contraction of the related muscles. Next, an anesthetic solution of Ropivacaine 0.375% (dose 37.5 mg) plus Mepivacaine 1% (dose 100 mg) and Dexamethasone 4mg, total volume 21 ml, will be injected.
  Lateral femoral cutaneous, femoral and obturator nerve blocks, femoral will be performed with the ultrasound technique. After identifying the nerves, a needle will be inserted with an "in plane" approach and will be injected.
  The anesthesia mixture will consist for all of :Ropivacaine 0.375% plus Mepivacaine 1% plus dexamethasone 4 mg.
  The volumes of the 3 anesthesia mixtures will be respectively: 1ml, 15ml,5ml.
  Arms: Peripheral nerve blocks
Drug: Anesthesiological mixtures (Spinal anesthesia) — The anesthesia mixtures will be injected into the subarachnoid space for spinal anesthesia. It will consist of the following local anesthetics and adjuvants: Hypobaric Bupivacaine 0.5% 7.5 mg and Sufentanil 5 µg.
  Arms: Selective Spinal Anesthesia
Drug: Anesthesiological mixtures (Peripheral nerve block) — The anesthesia mixtures will be injected into selected peripheral nerves . It will consist of the following local anesthetics and adjuvants: Ropivacaine 0.375% plus Mepivacaine 1% and Dexamethasone 4 mg.
  Arms: Peripheral nerve blocks

SUMMARY:
Proximal Femur Fractures (PFF) represent one of the most common orthopedic injuries worldwide, affecting especially elderly patients with potentially disabling outcomes and a marked impairment of quality of life. Taking into account their inherent instability, PFF are usually treated surgically within the shortest possible delay in order to reduce the risk of major and minor complications, the length of hospitalization and related costs. In this setting, most retrospective and prospective studies have reported a similar 30-day mortality rate comparing Spinal Anesthesia (SA) and General Anesthesia (GA), often recommending an adjuvant Peripheral Nerve Block (PNBs) to control postoperative pain. There is consensus that anticoagulant therapy, lack of pharmacological optimization or other conditions may represent a contraindication to SA. In these cases, blocking the nerves responsible for innervation of the proximal femur (i.e., the femoral, lateral femoral-cutaneous, obturators and sciatic nerves) may be a useful option. This study will aim to compare the incidence of intraoperative and postoperative adverse events, as well as the analgesic efficacy of the PNBs compared to SSA in patients diagnosed with PFF who underwent intramedullary nailing as a method of fixation.

DETAILED DESCRIPTION:
A venous access (16-18 G) will be placed in the operating room and antibiotic prophylaxis will be administered (Cefazolin 1 or 2 gr. iv or, in case of allergy, Clindamycin 600 mg iv). Pantoprazole 40 mg iv will also be administered. Pulse oximetry (SpO2), heart rate (HR), body temperature (C°), continuous invasive blood pressure (cIBP), brain oximetry with ForeSight will be monitored. Risk factors of Postoperative Nausea and Vomiting (PONV) will be assessed using the Apfel score. Antiemetic prophylaxis will be administered in accordance with the 2020 Fourth Consensus Guidelines for the Management of PONV. A pre-loading will be started with 500 ml of crystalloids iv will be administered; pre-procedural sedation will be performed with Midazolam 0.03 mg/Kg until a Richmond Agitation Sedation Scale (RASS) -1 or -2 will be obtained. All patients will receive intraoperative sedation with Dexmedetomidine 0.7 gamma/Kg/h and o2-therapy with a nasal cannula with a flow rate of 2L/min. We will also proceed to an intraoperative fluid administration of 15-20 ml / kg / hour of iv crystalloids. Rate of hypotension and bradycardia will be monitored during surgery. At this point, the type of anesthesia will be followed based on the randomization group.The following variables will be evaluated:

* intraoperative haemodynamic adverse events (rates of hypotension and bradycardia)
* postoperative adverse events (rates of nausea/vomiting and delirium and rate of deep vein thrombosis, myocardial infarction and neurological lesion during the hospital stay);
* postoperative pain evaluated by NRS and PAINED
* time to mobilization
* need of analgesic rescue dose after surgery
* lenght of stay
* bromage and hollmen scale of healthy limb and fractured limb assessed at different time
* surgical satisfaction (evaluated with 6-point Likert scale).
* the duration of surgery (min)

ELIGIBILITY:
"Inclusion Criteria" :

* Subject has signed and dated an Informed Consent Form
* Subject is classified as a ASA (American Society of Anesthesiologists) status I-IV
* Subject is age over 65 years old
* Subjects with femur fracture, candidates for intramedullary nailing surgery, to be operated on within 48 hours

"Exclusion Criteria":

* Age younger than 65 years
* Subject with contraindications to subarachnoid technique or peripherical nerve blocks
* Subject with local anesthetic allergy
* Subject in whom the treatment protocol could not be fully applied were excluded from this study.
* Study refusal
* Neurological disease of the lower limbs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain evaluated by NRS scales | Every 6 hours during treatment until the first 24 postoperative hours
  NRS assessment will be carried out using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". patients will be asked to circle the number between 0 and 10 that fits best to their pain intensity.
Postoperative pain evaluated by PAINAD scales | Every 6 hours during treatment until the first 24 postoperative hours
  The PAINED scale (Pain Assessment in Advanced Dementia Scale) assesses 5 items: facial expression, breathing, negative vocalizations, consolability and body language with a range from 0 to 10 (1-3=mild pain; 4-6=moderate pain; 7-10=severe pain).
Rate of postoperative nausea and vomiting (PONV) | Every 6 hours during treatment until the first 24 postoperative hours
  We will analyze the risk factors of postoperative nausea and vomiting (PONV) by administering an Apfel score to each patient, practicing intraoperative and postoperative antiemetic treatment in accordance with the 2020 Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting.
Rate of Delirium | Every 6 hours during treatment until the first 24 postoperative hours
  Postoperative delirium (POD) is an acute and fluctuating alteration of mental state of reduced awareness and disturbance of attention, which begins in the recovery room and occurs up to 5 days after surgery. POD will be detected by "3-Minute Diagnostic Confusion Assessment Method" (3D-CAM) and has four features: (1) altered mental status/fluctuating course, (2) inattention, (3) altered level of consciousness, and (4) disorganized thinking [27]. For the prevention and treatment of POD, we will follow the 2017 European Society of Anesthesiology guidelines.
Rate of deep vein thrombosis | up to 1 weeks
  The diagnosis of Deep Vein Thrombosis will be based on postoperative observations of the affected limbs during the patient's hospital stay; the following manifestations will be monitored: limb swelling, pain, elevated skin temperature, changes in skin color, venous return disorders, Homans' sign, and Neuhof's sign. Color-Doppler ultrasound will be performed bilaterally, in case of positivity of clinical signs and symptoms.
Rate of myocardial infarction | up to 1 weeks
  The typical symptoms of myocardial ischemia, combined with characteristic changes on an ECG and a significant increase in blood levels of high-sensitivity cardiac troponins, will be used to diagnose a Myocardial Infarction. In cases where the diagnosis is uncertain, it will be necessary to conduct additional non-invasive evaluations, such as an echocardiogram
Rate of neurological lesion | up to 1 weeks
  Neurological lesion was evaluated based on the presence of sensory, motor, or both neurological symptoms
Intraoperative haemodynamic adverse events | From the beginning to the end of surgery
  Hypotension defined as a Systolic Blood Pressure (SBP) of less than 90 mm Hg for more than 5 minutes or a decrease of 35% in the Mean Arterial Pressure (MAP). Bradicardia, indicated by a heart rate of fewer than 60 beats per minute for more than 5 minutes.

SECONDARY OUTCOMES:
Need of analgesic rescue dose | From the end of treatment to 24 hours postoperatively
  time between anesthesia and first analgesic rescue dose.Pharmacological therapy will be based on the patients' responses. After surgery, we will administer intravenous paracetamol 1 g 3 times a day. Ketorolac 30 mg (not for glomerular filtration rate < 50 ml/min) or Oxycodone (up to 0.1mg/Kg) mg will be available as rescue dose. Pain control will be considered good in case of NRS and PAINED score less than or equal to 4.
Time to mobilization (hours) | Time to mobilization will be assessed immediately after the locoregional procedure, up to 24 hours postoperatively.
  Time to mobilization (hours), defined as the time (hours) between LA injection and lower limb mobilization (score 4) on the Bromage scale (1, unable to move feet or knees; 2, able to move feet only; 3, just able to move knees; 4, full flexion of knees and feet).
Lenght of stay (days) | from date of hospital admission up to 1 weeks
  Lenght of stay (days), defined as days from hospital admission to discharge, will be reported.
Bromage and Hollmen scale of healthy limb and fractured limb assessed at different time | Motor block and sensory block were assessed before LA injection (baseline time) and 10 , 15 and 20 minutes after baseline time and every 30 minute during the surgery
  During the execution of the anesthesiologic procedures, the motor and sensory blocks will be tested bilaterally using the "Bromage scale" and with the "Hollmen scale", respectively. The presence of complete motor block (Bromage 1) with "unable to move feet or knees", and complete sensory block (Hollmen 4), tested by pinprick and ice test, defined as "loss of sensation" in the affected limb, will define an adequate anesthesiological plane.

OTHER OUTCOMES:
The duration of surgery (min) | From the beginning of surgery up to 120 minutes
  The duration of surgery (min), assessed as Planned time(min) and Effective time(min)
Surgical satisfaction related to anesthesiological plane | 1 hours after surgery
  will be obtained with a 6-point Likert scale score filled out by the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Coviello, Researcher, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coviello A, Cirillo D, Bernasconi A, de Siena AU, Spasari E, Barone MS, Piccione I, Ranieri G, Tognu A, Servillo G, Iacovazzo C. Peripheral nerve blocks vs selective spinal anesthesia in patients with femur fracture: a patient-, surgeon-, and assessor-blinded randomized controlled study. J Anesth Analg Crit Care. 2025 Dec 3;5(1):88. doi: 10.1186/s44158-025-00302-6. PMID 41340155